CLINICAL TRIAL: NCT04661956
Title: The Diagnostic Yield and Safety of Transbronchial Cryobiopsy Under The Guidance of The Endobronchial Ultrasound in The Pulmonary Periphral Nodule: A Multicenter Prospective Random Control Trial
Brief Title: The Diagnostic Yield and Safety of Transbronchial Cryobiopsy in The Pulmonary Periphral Nodule
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ShiYue Li (Other)
Responsible Party: Sponsor-Investigator, ShiYue Li, Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20200914
Record Dates: First submitted 2020-10-26; First posted 2020-12-10 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Diagnosis; Complication Rate
Keywords: Transbronchial Cryobiopsy; Diagnostic Yield; Safety; Pulmonary Periphral Nodule
MeSH Terms: conditions — Disease | interventions — Surgical Instruments

STUDY DESIGN:
Intervention Model Description: a prospective multicenter random control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transbronchial cryobiopsy (Experimental): Transbronchial cryobiopsy was performed in the patiens of pulmonary peripheral nodule
  Interventions: Procedure: Transbronchial cryobiopsy/Transbronchial lung biopsy (forcep)
- Transbronchial lung biopsy (Other): Transbronchial lung biopsy was performed in the patiens of pulmonary peripheral nodule
  Interventions: Procedure: Transbronchial cryobiopsy/Transbronchial lung biopsy (forcep)

INTERVENTIONS:
Procedure: Transbronchial cryobiopsy/Transbronchial lung biopsy (forcep) — Transbronchial lung biopsy by cryoprobe or by forcep

SUMMARY:
Transbronchial cryobiopsy under the guidance of endobronchial ultrasound is performed in patients with pulmonary peripheral nodule, and assess the diagnostic yield and safety.

DETAILED DESCRIPTION:
Transbronchial cryobiopsy under the guidance of endobronchial ultrasound is performed in patients with pulmonary peripheral nodule, and assess the diagnostic yield and safety. This is a multi-center prospective randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

1. The patients are admitted as Pulmonary Periphral Nodule, while undefined after thorough history collection, laboratory examination and radiological data.
2. The longest diameter of the Pulmonary Periphral Nodule is less than 30mm in HRCT.
3. The Pulmonary Periphral Nodule can be detected by radial-EBUS
4. Transbronchial cryobiopsy(TBCB) is indicated by clinicians for definitive diagnosis and patients are content with the examination with agreement signed.
5. Routine blood test, ECG examination, coagulation function, chest HRCT have been completed.

Exclusion Criteria:

1. The longest diameter of the Pulmonary Periphral Nodule is more than 30mm.
2. The Pulmonary Periphral lesions cannot be detected by the radial endobronchial ultrasound.
3. The clinical examinations mentioned above are not completed. The patient cannot endure or does not agree the procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Diagnotic yield | six months
  Percentage of definitive pathological diagnosis by transbronchial cryobiopsy

SECONDARY OUTCOMES:
Complication rate | one week
  Incidence of bleeding, pneumothorax (during the procedure and within 7 days after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, master, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (24):
- China (24):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - AnHui Chest Hospital, Hefei, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Xiamen Second Hospital, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen Guangming New District People's Hospital, Shenzhen, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Central Hospital Of WuHan, Wuhan, Hubei
  - Hubei Provincial Hospital of Integrated Chinese & Western Medicine, Wuhan, Hubei
  - People's Hospital of Hunan Province, Changsha, Hunan
  - XiangYa Hospital Central South University, Changsha, Hunan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Xi'an chest hospital, Xi’an, Shanxi
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Zhejiang Provincial People' s Hospital, Huangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang